CLINICAL TRIAL: NCT00088998
Title: Phase II Trial Of Docetaxel With Capecitabine And Bevacizumab As First-Line Chemotherapy For Patients With Metastatic Breast Cancer
Brief Title: Docetaxel, Capecitabine, and Bevacizumab in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0432; NCI-2012-02617 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000377886 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Bevacizumab; Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + bevacizumab + capecitabine (Experimental): Patients receive docetaxel IV over 1 hour and bevacizumab IV over 30-90 minutes on day 1. Patients also receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive at least 2 additional courses beyond CR.
  Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: docetaxel

INTERVENTIONS:
Biological: bevacizumab
Drug: capecitabine
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as bevacizumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Bevacizumab may also stop the growth of tumor cells by stopping blood flow to the tumor. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel and capecitabine together with bevacizumab works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with metastatic breast cancer treated with docetaxel, capecitabine, and bevacizumab as first-line chemotherapy.

Secondary

* Determine time to disease progression in patients treated with this regimen.
* Determine survival of patients treated with this regimen.
* Determine the toxicity profile of this regimen in these patients.
* Determine the duration of response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour and bevacizumab IV over 30-90 minutes on day 1. Patients also receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive at least 2 additional courses beyond CR.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer

  * Clinical evidence of metastatic disease

    * No bone metastases as the only evidence of metastasis
* Measurable disease

  * At least 1 lesion ≥ 2.0 cm by CT scan or MRI OR ≥ 1.0 cm by spiral CT scan

    * Lesions on chest x-ray allowed provided they are clearly defined and surrounded by aerated lung
  * Clincal lesions only considered measurable when they are superficial (e.g., skin nodules or palpable lymph nodes)
  * Target lesion must not have been exposed to prior radiotherapy unless disease has progressed since completion of radiotherapy
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis or pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No HER2/neu-positive tumors by immunohistochemistry or amplified fluorescence in situ hybridization unless disease has progressed after trastuzumab (Herceptin®)-containing therapy alone or with antiestrogen hormonal therapy for metastatic disease OR trastuzumab is contraindicated
* Prior breast cancer allowed
* No prior or active brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* No bleeding diathesis or uncontrolled coagulopathy

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * AST and ALT normal AND alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
  * AST and ALT ≤ 1.5 times ULN AND alkaline phosphatase ≤ 2.5 times ULN
  * AST and ALT ≤ 5 times ULN AND alkaline phosphatase normal

Renal

* Creatinine clearance ≥ 30 mL/min
* No proteinuria OR
* Protein < 1 g by 24-hour urine collection
* No nephrotic syndrome

Cardiovascular

* No uncontrolled hypertension (i.e., blood pressure > 160/90 mm Hg on ≥ 2 different observations ≥ 5 minutes apart)

  * Blood pressure < 140/90 mm Hg on ≥ 3 different observations over ≥ 14 days, for patients who recently began or adjusted anti-hypertensive medication
* No atrial or venous thrombosis within the past month
* No clinically significant heart disease, including any of the following:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Uncontrolled cardiac arrhythmias
  * Unstable angina
* No myocardial infarction within the past 12 months
* No history of cerebrovascular accident

Pulmonary

* No hemoptysis within the past 6 months

Gastrointestinal

* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome
* Able to receive oral medication

Other

* No other stage III or IV invasive malignancy requiring treatment within the past 5 years
* No pre-existing peripheral neuropathy > grade 1
* No history of allergy or hypersensitivity to study drugs, agents that are chemically similar to study drugs, or drugs that contain polysorbate 80
* No prior severe reaction to fluoropyrimidines
* No known hypersensitivity to fluorouracil
* No known dihydropyrimidine dehydrogenase deficiency
* No active infection
* No significant medical condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No other concurrent biologic therapy

Chemotherapy

* Prior adjuvant or neoadjuvant chemotherapy allowed for primary disease
* No prior chemotherapy for metastatic disease
* More than 4 weeks since prior cytotoxic chemotherapy
* More than 6 months since prior taxanes (e.g., docetaxel or paclitaxel)
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* Prior antiestrogen hormonal therapy allowed in the adjuvant or metastatic setting

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy to a target lesion

  * Prior single-dose palliative radiotherapy allowed within the past 4 weeks
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery

Other

* More than 2 weeks since prior aspirin, anticoagulants, or thrombolytic agents

  * Concurrent low-dose warfarin (1 mg/day) to maintain patency of vascular access device allowed
* More than 4 weeks since prior investigational agents
* No concurrent aspirin, anticoagulants, or thrombolytic agents
* No concurrent participation in another clinical trial involving investigational agents or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-12; Primary Completion 2006-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response (complete or partial) rate as measured by RECIST | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Perez EA, Hillman DW, Dentchev T, Le-Lindqwister NA, Geeraerts LH, Fitch TR, Liu H, Graham DL, Kahanic SP, Gross HM, Patel TA, Palmieri FM, Dueck AC. North Central Cancer Treatment Group (NCCTG) N0432: phase II trial of docetaxel with capecitabine and bevacizumab as first-line chemotherapy for patients with metastatic breast cancer. Ann Oncol. 2010 Feb;21(2):269-274. doi: 10.1093/annonc/mdp512. Epub 2009 Nov 9. PMID 19901014